CLINICAL TRIAL: NCT00133341
Title: Clinical Evaluation of the 3 Allergens: Methyldibromoglutharonitrile, Parthenolide and Goldnatriumthiosulphate for "TRUE Test® Panel 3" - a Phase II, Dose-Response Study.
Brief Title: Clinical Evaluation of the 3 Allergens: Methyldibromoglutharonitrile, Parthenolide and Goldnatriumthiosulphate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mekos Laboratories AS (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: MEKOS 05 P379/1
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2006-02-27 (Estimated); Status verified 2006-02

CONDITIONS: Allergic Contact Dermatitis
Keywords: Allergic contact dermatitis,patch testing, dilution series
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — 1,2-dibromo-2,4-dicyanobutane; parthenolide

INTERVENTIONS:
Drug: Goldnatriomthiosulphate, MDBGN, parthenolide

SUMMARY:
It is the purpose of this study to determine the concentration of 3 allergens (goldnatriumthiosulphate, methyldibromoglutharonitrile [MDBGN], parthenolide) for diagnosing allergic contact dermatitis.

DETAILED DESCRIPTION:
The TRUE Test standard panel consists of two tape strips, panel 1 with 11 allergen patches and a negative control and panel 2, with 12 allergen patches. TRUE test panel 1 and 2 contain 23 of the most frequent contact allergens.With these 23 allergens, it is possible to detect about 60-70% of contact allergic reactions. Thus, there is a need for expanding the number of allergens included in TRUE Test in order to detect more contact allergic reactions. Therefore goldnatriumthiosulphate, methyldibromoglutharonitrile and parthenolide are developed for inclusion in a third TRUE Test panel. This study is a dose-response study using 3 dilution series to detect the optimum concentration of the 3 allergens. A phase-III study will be performed afterwards to establish the efficacy and safety of the three allergens.

ELIGIBILITY:
Inclusion Criteria:

* Positive MDBGN patch test within the latest 5 years or positive Parthenolide patch test within the latest 5 years or positive Goldnatriumthiosulphate patch test within the latest 5 years.
* Age more or equal to 18 years.
* Signed informed consent.

Exclusion Criteria:

* Topical treatment with corticosteroids or immunosuppressives during the latest 7 days on the test area or near the test area.
* Systemic treatment with corticosteroids or immunosuppressives during the latest 7 days.
* Treatment with UV-light during the latest 3 weeks.
* Widespread active dermatitis or dermatitis on test area.
* Breast-feeding, pregnancy or insufficient contraception. If any doubt a negative urine-pregnancy test should be demonstrated or the patch test should be postponed one period.
* Subjects not able to cooperate.
* Participation in other clinical studies during the study period and 3 weeks prior to study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-04; Study Completion 2005-12

PRIMARY OUTCOMES:
Skin reaction from the 3 patch tests. (Allergic or irritant reaction, grade)

SECONDARY OUTCOMES:
Vehicle (polyvinylpyrrolidone [PVP] or hydroxypropylcellulose [HPC])

CONTACTS AND LOCATIONS:
Overall Officials: Klaus E Andersen, Prof., Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Odense C, Denmark